CLINICAL TRIAL: NCT02579018
Title: Heart Rate Sensing and Response in Persons With Anorexia Nervosa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: Pro00064421
Record Dates: First submitted 2015-10-15; First posted 2015-10-19 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-12

CONDITIONS: Anorexia Nervosa
Keywords: Anorexia Nervosa; Exercise; Healthy Adults; Physical Activity
MeSH Terms: conditions — Anorexia Nervosa; Motor Activity

ARMS (3):
- Anorexia Nervosa (AN) (Experimental): Diagnosis of anorexia spectrum disorder and stable use of all medications ≥ three months.
  Interventions: Behavioral: One hour supervised exercise session
- Matched Controls (Experimental): No diagnosis of anorexia spectrum disorder. Stable use of all medications ≥ three months. Also age (+/- 2 years) and gender matched to AN study participant and exercise regularly.
  Interventions: Behavioral: One hour supervised exercise session
- Healthy Controls (Experimental): No diagnosis of anorexia spectrum disorder. Stable use of all medications ≥ three months. Do not exercise regularly.
  Interventions: Behavioral: One hour supervised exercise session

INTERVENTIONS:
Behavioral: One hour supervised exercise session — All participants will participate in a one hour supervised exercise session. Participants will wear a physical activity monitor during the assessment for continuous monitoring of heart rate. Short, intense bouts of exercise will be interspersed with rest periods.

SUMMARY:
There are two major goals of this investigation. First, to develop pilot data to justify a larger randomized clinical trial of an intervention designed to train interoceptive signals (IS) and interoceptive responsivity (IR) in persons with Anorexia Nervosa (AN). Second, the investigators will determine whether persons with AN have similar or different IS and IR for heart rate while exercising as compared to age and gender matched controls.

DETAILED DESCRIPTION:
The purpose of this pilot investigation is to assess AN interoceptive sensitivity and responsivity as it pertains to heart rate during exercise. Thirty adults, 18 years and older will be recruited for a cross-sectional comparison of IS and IR in the context of exercise.

ELIGIBILITY:
Inclusion Criteria: Study participants will include adults with anorexia spectrum disorders and healthy age and gender matched controls. There will be two control groups, one that includes regularly exercising age and gender matched persons and one where controls do not engage in regular exercise.

For those with AN, the following INCLUSION criteria must be met:

* Age ≥ 18 years old
* BMI 25 kg/m2 or less
* Diagnosis of anorexia spectrum disorder
* Medications: Stable use of all medications ≥ three months

For age and gender matched controls, the following INCLUSION criteria must be met:

* Age ≥ 18 years old
* BMI 25 kg/m2 or less
* No diagnosis of anorexia spectrum disorder
* Medications: Stable use of all medications ≥ three months
* Age (+/- 2 years) and gender matched to study participant

Exclusion Criteria:

* History of diabetes, heart disease or taking medications for those conditions
* History of hypertension (high blood pressure) not controlled with medication
* Orthopedic limitations, musculoskeletal disease and/or injury
* Inability to consent
* Lack of transportation to the Duke Center for Living campus

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-03; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Mean percentage of time in prescribed heart rate range during four bouts of interval exercise training | Baseline only
  One exercise training session

CONTACTS AND LOCATIONS:
Overall Officials: Nancy L Zucker, PhD, Principal Investigator — Director, Duke Center for Eating Disorders
Locations (1):
- Duke Medicine - Duke Molecular Physiology Institute, Durham, North Carolina, United States